CLINICAL TRIAL: NCT02649621
Title: The Effect of in Vivo Cultured Limbal Stem Cells in the Treatment of Unilateral Corneal Stem Cell Damage
Brief Title: The Improvement of Limbal Stem Cell Deficiency (LSCD) in Unilateral Stem Cell Damage by Amniotic Membrane Extract Eye Drop (AMEED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Eye-002
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Limbal Stem Cell Deficiency (LSCD)
Keywords: Limbal Stem Cell Deficiency Amniotic Membrane Extract Eye Drop in vivo cultivation
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amniotic Membrane Extract Eye Drop recipient (Experimental): patients with limbal stem cell Deficiency who receive amniotic membrane transplantation and amniotic membrane extract eye drop as eye drop.
  Interventions: Biological: Amniotic Membrane Extract Eye Drop (AMEED)

INTERVENTIONS:
Biological: Amniotic Membrane Extract Eye Drop (AMEED) — Use of use Amniotic Membrane Extract Eye Drop (AMEED) on in vivo cultured limbal stem cells in the treatment of unilateral corneal stem cell damage.

SUMMARY:
Corneal epithelial cells and limbal stem cells (LSC) are located in the limbus basal epithelium that are necessary for repair of corneal. About patients with deficient or absence of this area has been proposed various treatments such as limbal stem cell transplantation.

This study is a prospective clinical trial to compare the improvement of limbal stem cell deficiency (LSCD) in vivo by using of Amniotic Membrane Extract Eye Drop (AMEED).

DETAILED DESCRIPTION:
The cornea is the eye anterior portion which its refractive power and transparent is essential for normal vision.

The damaged cornea surface can reduce vision and leads to blindness, ultimately. Corneal epithelial and some times, limbal stem cell (LSC) are involved in corneal injuries. Limbal stem cells (LSC) are necessary for repair and reconstruction of corneal that reduction of these cells occurs by various causes including congenital causes, eye inflammatory diseases and burns. For cornea stem cell damages or limbal stem cell deficiency (LSCD), cornea becomes conjunctivalization. LSCD may involve one eye (unilateral) or two eyes (bilateral).

Due to autologous transplantation problems in patients with unilateral LSCD and recent successes to resolve this problem, it seems that transplantation of cultured corneal stem cells on amniotic membrane is other way in treatment of unilateral LSCD. It is called ex vivo.

Amniotic membrane can modulate corneal epithelium healing by promoting re-epithelialization and migration of limbal stem cell while suppressing stromal inflammation, angiogenesis and scarring. It is well accepted that amniotic membrane transplantation (AMT) as a temporary patch normally dissolves within 2 weeks. Consequent reapplication of membrane is difficult for the patient. On the other hand, in ex vivo, corneal tissue from healthy eye must be transported to laboratory for cell culture on AM that is required equipment. There is, also, a risk of cell infection and transmission that is very important issue. However, in infected cells, re-biopsy of the healthy eye is required that is uncomfortable and difficult for the patient. Other studies have been reported that amniotic membrane extract (AME) has same characteristics and features.

We previously have reported an effective potential of AMEED in limbal stem cell proliferation in vitro and also rabbit corneal epithelium healing in vivo.

This study is a prospective clinical trial to use Amniotic Membrane Extract Eye Drop (AMEED) on in vivo cultured limbal stem cells in the treatment of unilateral corneal stem cell damage.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unilateral chemical burn (grade III to up); estimation of chemical burns amount and classification was according to Dua.
* Without Age limitation

Exclusion Criteria:

* Lack of timely referral of patients for examinations
* Simultaneous use of other drugs that cause impairment of the data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Limbal defect size | 12 months
  The measurement of limbal defect size by microscope 12 months after corneal surgery
Corneal epithelial integrity | 12 months
  The measurement of Corneal epithelial integrity by microscope 12 months after corneal surgery
Corneal epithelial stability | 12 months
  The measurement of Corneal epithelial stability by microscope 12 months after corneal surgery

SECONDARY OUTCOMES:
Vascularization | 12 months
  Evaluation the rate of corneal vascularization with microscope 12 months after surgery.
Transparency | 12 months
  Evaluation the transparency with visual tests 12 months after surgery.
Best spectacle corrected visual activity | 12 months
  Evaluation the best spectacle corrected visual activity with visual tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Marzieh Ebrahimi, PhD, Study Director — Department of Regenerative Biomedicine at Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Alireza Baradaran, MD, Study Director — Labafi Nejad Eye Research Center, Tehran, Iran; Mitra Akbari, MD, Principal Investigator — Labafi Nejad Eye Research Center, Tehran, Iran; Niloufar Shayan, MSc, Principal Investigator — Department of Stem Cells and Developmental Biology at Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Maryam Momeni, MSc, Principal Investigator — Department of Stem Cells and Developmental Biology at Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://royaninstitute.org